CLINICAL TRIAL: NCT07027176
Title: Effects of Walking Exercise on Sleep Quality, Memory, and Attention in Older Adults With Poor Sleep Quality
Brief Title: Effects of Walking Exercise on Sleep Quality in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yea-Ru Yang (Other)
Responsible Party: Sponsor-Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Organization: National Yang Ming Chiao Tung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU114071AF
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Sleep Quality; Cognitive Function
Keywords: sleep quality; physical activity; memory; attention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- low-intensity exercise in the morning (Experimental)
  Interventions: Behavioral: walking exercise
- moderate-intensity exercise in the morning (Experimental)
  Interventions: Behavioral: walking exercise
- low-intensity exercise at night (Experimental)
  Interventions: Behavioral: walking exercise
- moderate-intensity exercise at night (Experimental)
  Interventions: Behavioral: walking exercise
- control group (No Intervention)

INTERVENTIONS:
Behavioral: walking exercise — Divided into low-intensity and moderate-intensity exercise intervention groups, participants exercised either during the day or at night. The intervention lasted for 12 weeks.
  Arms: low-intensity exercise at night; low-intensity exercise in the morning; moderate-intensity exercise at night; moderate-intensity exercise in the morning

SUMMARY:
This study aims to explore whether increasing physical activity can improve sleep quality in older adults, particularly those with poor sleep, and whether such improvements positively influence cognitive functions such as memory and attention. The goal is to provide a practical intervention strategy to enhance both sleep quality and cognitive function, contributing to healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60 and 80
* Montreal Cognitive Assessment score > 26
* Pittsburgh Sleep Quality Index score > 5
* Not participated in any regular exercise program in the past 3 months
* Being able to understand and follow the exercise program

Exclusion Criteria:

* Suffering from any neurological or musculoskeletal disorders
* Visual problems
* Geriatric Depression Scale score ≥ 6
* Vestibular disease or vestibular dysfunction
* Being unable to walk independently due to neuromuscular or musculoskeletal limitations
* A history of mental illness
* Untreated obstructive sleep apnea
* A history of electroconvulsive therapy or severe head injury leading to prolonged unconsciousness
* A history of alcoholism or dependence within the past 2 years
* A history of cancer within the past 5 years
* Any major systemic diseases, unstable medical conditions (such as insulin-dependent diabetes or uncontrolled diabetes, uncontrolled hypertension (systolic pressure > 170 or diastolic pressure > 100 mmHg)),
* Taking medications that affect the central nervous system, balance, coordination, or sleep (such as antidepressants, vestibular sedatives or anxiolytics, sleep aids)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Chinese version of the Pittsburgh Sleep Quality Index | From pre-intervention to the end of intervention at 12 weeks
  sleep quality
Digital Span Test | From pre-intervention to the end of intervention at 12 weeks
  short-term memory and attention
Chinese version Verbal Learning Test | From pre-intervention to the end of intervention at 12 weeks
  short-term memory
Chinese Version Trail Making Test | From pre-intervention to the end of intervention at 12 weeks
  attention
Chinese version of Stroop Color and Word test | From pre-intervention to the end of intervention at 12 weeks
  attention

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | From pre-intervention to the end of intervention at 12 weeks
  general cognitive function
Six-Minute Walk Test | From pre-intervention to the end of intervention at 12 weeks
  walking endurance
Multidimensional Fatigue Inventory | From pre-intervention to the end of intervention at 12 weeks
  fatigue condition
Depression Anxiety Stress Scales-21 | From pre-intervention to the end of intervention at 12 weeks
  depression, anxiety and stress condition
Heart rate variability | From pre-intervention to the end of intervention at 12 weeks
  autonomic nervous system function

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Assistive Technology, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No